CLINICAL TRIAL: NCT05382312
Title: A Parallel Group, Phase 2A, Randomised, Open Label Treatment Study to Assess the Early Bactericidal Activity, Safety and Tolerability of GSK3036656 Administered as a Two Drug Combination With Novel and Established Antitubercular Agents, or Standard of Care in Adults With Rifampicin-susceptible Pulmonary Tuberculosis
Brief Title: Early Bactericidal Activity, Safety & Tolerability of Oral GSK3036656 in a Dual Combination With Novel and Established Antitubercular Agents, or Standard of Care in Adults With Rifampicin Susceptible Pulmonary Tuberculosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: Click-TB Consortium (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 214912
Record Dates: First submitted 2022-05-16; First posted 2022-05-19 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-09

CONDITIONS: Tuberculosis
Keywords: Early bactericidal activity; Pulmonary tuberculosis; RIFAFOUR; Bedaquiline; Delamanid; GSK3036656; BTZ-043
MeSH Terms: conditions — Tuberculosis; Tuberculosis, Pulmonary | interventions — GSK656; bedaquiline; OPC-67683; 2-(2-methyl-1,4-dioxa-8-azaspiro(4.5)dec-8-yl)-8-nitro-6-(trifluoromethyl)-4H-1,3-benzothiazin-4-one

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: All laboratory staff involved in analyzing and reporting the microbiological endpoints (logarithm to base10 [log10] colony forming units [CFU] counts and time to sputum culture positivity) will be unaware of treatment assignments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Participants receiving GSK3036656+bedaquiline (Experimental)
  Interventions: Drug: GSK3036656; Drug: Bedaquiline
- Participants receiving GSK3036656+delamanid (Experimental)
  Interventions: Drug: GSK3036656; Drug: Delamanid
- Participants receiving bedaquiline+delamanid (Experimental)
  Interventions: Drug: Bedaquiline; Drug: Delamanid
- Participants receiving RIFAFOUR e-275 (Experimental)
  Interventions: Drug: RIFAFOUR e-275
- Participants receiving GSK3036656+BTZ-043 (Experimental)
  Interventions: Drug: GSK3036656; Drug: BTZ-043

INTERVENTIONS:
Drug: GSK3036656 — GSK3036656 will be administered.
  Arms: Participants receiving GSK3036656+BTZ-043; Participants receiving GSK3036656+bedaquiline; Participants receiving GSK3036656+delamanid
Drug: Bedaquiline — Bedaquiline will be administered.
  Arms: Participants receiving GSK3036656+bedaquiline; Participants receiving bedaquiline+delamanid
Drug: Delamanid — Delamanid will be administered.
  Arms: Participants receiving GSK3036656+delamanid; Participants receiving bedaquiline+delamanid
Drug: RIFAFOUR e-275 — RIFAFOUR e-275 will be administered.
  Arms: Participants receiving RIFAFOUR e-275
Drug: BTZ-043 — BTZ-043 will be administered.
  Arms: Participants receiving GSK3036656+BTZ-043

SUMMARY:
This study aims to measure the early bactericidal activity (EBA), safety, tolerability and pharmacokinetics with GSK3036656 in combination with either delamanid or bedaquiline or BTZ-043, delamanid in combination with bedaquiline or standard of care for 14 days in participants with newly diagnosed sputum smear positive drug-sensitive pulmonary tuberculosis. Participants will revert to the standard treatment (RIFAFOUR® e-275) once the study treatment (Day 1 to Day 14) has been completed.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be 18 to 65 years of age inclusive, at the time of signing the informed consent.
* Participants who have:

  1. New episode of untreated, rifampicin-susceptible pulmonary tuberculosis (TB)
  2. A chest X-ray picture consistent with pulmonary TB
  3. At least one sputum sample positive on direct microscopy for acid-fast bacilli (at least 1+ on the International Union Against Tuberculosis and Lung Disease [IUATLD]/World Health Organization [WHO] scale) or positive on a molecular test (at least medium positive for MTB on Xpert MTB/Rif)
  4. Normal echocardiogram or echocardiogram with normal left ventricular function with at most trace to mild valvular regurgitation is allowed and no valvular stenosis.
  5. A creatinine clearance greater than or equal to (>=)90 mL/minute (Cockroft-Gault formula).
* Male participants are eligible to participate if they agree to barrier precautions until 90 days after last dose.
* A female participant is eligible to participate if she is not pregnant or breast feeding and is a woman of non-childbearing potential (WONCBP) or a woman of childbearing potential (WOCBP) using a contraceptive method that is highly effective. A WOCBP must have a negative pregnancy test urine or serum as required by local regulations before the first dose of study intervention. Only participants who are at least 25 years of age (and females of non-childbearing potential) will be eligible for the positron emission tomography-computed tomography (PET-CT) assessments.
* Capable of giving signed informed consent.

Exclusion Criteria:

* Evidence of a clinically significant (as judged by the Investigator) condition or abnormality (other than the indication being studied) that might compromise safety or the interpretation of trial efficacy or safety endpoints.
* Clinically significant evidence of extrathoracic TB as judged by the Investigator.
* QTc interval corrected for heart rate by Fridericia's formula (QTcF) greater than (>)450 milliseconds (msec).
* Arterial hypertension with Systolic BP >=160 mm Hg or diastolic BP >=100 nm Hg. Participants with well-controlled hypertension may be included if they are using amlodipine for the duration of the study.
* Participants with vitiligo.
* Participants receiving any QT prolonging drugs, including but not limited to fluoroquinolones, macrolides and clofazimine.
* HIV infected participants:

  1. having a cluster of differentiation (CD)4+ count <350 cells/microliters;
  2. having received any antiretroviral therapy medication within the last 30 days;
  3. or having received oral or intravenous antifungal medication within the last 30 days;
  4. or with an acquired immunodeficiency syndrome (AIDS)-defining opportunistic infection or malignancies in the last 12 months (except pulmonary TB).
* Presence of Hepatitis B surface antigen (HBsAg) or Positive Hepatitis C antibody test result at screening.
* Participants with diabetes (Type 1 or 2), point of care glycated hemoglobin (HbA1c) above 6.5%, or random glucose over 11.1 millimoles (mmol)/L
* Any diseases or conditions in which use of delamanid or bedaquiline is contraindicated.
* Participants with abnormal laboratory values at screening as graded by the enhanced Common Terminology Criteria for Adverse Events (CTCAE version 5 2017).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2022-07-26 (Actual); Primary Completion 2025-05-27 (Actual); Study Completion 2025-05-27 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in log10 CFU of Mycobacterium tuberculosis (MTB) (per milliliters of respiratory sputum samples) | Baseline and up to Day 14
  The extended early bactericidal activity of each treatment group will be determined by the change from Baseline to Day 14 in log10CFU.

SECONDARY OUTCOMES:
Change from Baseline in time to sputum culture positivity | Baseline and up to Day 14
  Time to sputum-culture positivity is the time between sample inoculation and detection of mycobacterial growth in the mycobacterium growth indicator tube.
Number of participants with serious adverse events | Up to Day 28
Number of participants with adverse events of Grade 3 severity or higher | Up to Day 28
Number of participants with adverse events related to study drug | Up to Day 28
Number of participants withdrawn from the treatment due to adverse events | Up to Day 28
Number of participants withdrawn from the study due to adverse events | Up to Day 28
Number of participants with electrocardiogram (ECG) values of potential clinical importance (PCI) | Up to Day 28
Number of participants with hematology laboratory values of PCI | Up to Day 28
Number of participants with clinical chemistry laboratory values of PCI | Up to Day 28
Number of participants with vital signs of PCI | Up to Day 28

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Bellville, South Africa

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.